CLINICAL TRIAL: NCT01315678
Title: Randomized, Open-Label, Active-Controlled, Multicenter Study to Assess the Efficacy, Safety and Tolerability of Arikayce™ in Cystic Fibrosis Patients With Chronic Infection Due to Pseudomonas Aeruginosa
Brief Title: Study to Evaluate Arikayce™ in CF Patients With Chronic Pseudomonas Aeruginosa Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR02-108
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: Pseudomonas Aeruginosa Infection
Keywords: Cystic Fibrosis; Respiratory Infections; Pulmonary Cystic Fibrosis; CFTR; Amikacin; Anti-bacterial Agents; Amikacin liposome inhalation suspension (ALIS)
MeSH Terms: conditions — Pseudomonas Infections; Cystic Fibrosis; Respiratory Tract Infections | interventions — Inhalation; Nebulizers and Vaporizers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arikayce™ (Experimental): Arikayce™ is liposomal amikacin for inhalation
  Interventions: Drug: Liposomal amikacin for inhalation (Arikayce™) using the PARI Investigational eFlow® Nebulizer.
- TOBI® (Active Comparator): TOBI® is tobramycin inhalation solution
  Interventions: Drug: Tobramycin inhalation solution using a PARI LC® Plus nebulizer.

INTERVENTIONS:
Drug: Liposomal amikacin for inhalation (Arikayce™) using the PARI Investigational eFlow® Nebulizer. — Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * liposomal amikacin for inhalation will be administered for 3 cycles where each cycle consists of 28 days on-treatment followed by 28 days off-treatment.
  Arms: Arikayce™
Drug: Tobramycin inhalation solution using a PARI LC® Plus nebulizer. — 300 mg tobramycin inhalation solution is administered twice a day using a PARI LC® Plus nebulizer.
  * Nebulization time is approximately 20 minutes for each administration.
  * Tobramycin inhalation solution will be administered for 3 cycles where each cycle consists of 28 days on-treatment followed by 28 days off-treatment
  Arms: TOBI®

SUMMARY:
A major factor in the respiratory health of Cystic Fibrosis (CF) participants is the prevalence of chronic Pseudomonas aeruginosa (Pa) infections. The Pa infection rate in CF patients increases with age and by age 18 years approximately 85% of CF patients in the US are infected. Liposomal amikacin for inhalation (Arikayce™) was developed as a possible treatment for chronic infection due to Pa in CF patients.

The purpose of this study is to determine whether Arikayce™ is effective in treating chronic lung infections caused by Pa in CF participants. The effectiveness, safety, and tolerability of Arikayce™ will be compared to Tobramycin TOBI®, an inhalation antibiotic already available for use.

DETAILED DESCRIPTION:
CF is a genetic disease resulting from mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene. Patients with CF manifest pathological changes in a variety of organs that express CFTR. The lungs are frequently affected often resulting in chronic infections by bacteria such as Pseudomonas aeruginosa and airway inflammation. Treatment of chronic lung infections is one of the principal goals of CF therapy. Arikayce™ LAI (liposomal amikacin for inhalation) is a sustained-release formulation of amikacin encapsulated inside nanoscale liposomal carriers designed for administration via inhalation. It is hypothesized that the sustained-release pulmonary targeting and biofilm penetration properties of this formulation will have several advantages over current therapies in treating CF patients with chronic lung infection caused by Pseudomonas aeruginosa.

This Phase 3 study has been designed to evaluate the efficacy, safety and tolerability of Arikayce™ in treating CF patients with chronic bronchopulmonary infection compared to a currently available antibiotic, TOBI® Inhalation Solution. Eligible participants will be randomized 1:1 to receive 590 mg of Arikayce™ once daily via a PARI Investigational eFlow® Nebulizer or 300 mg TOBI® BID via a PARI LC® PLUS nebulizer. Participants will receive 3 cycles of treatment with each cycle being comprised of 28 days on treatment followed by 28 days off-treatment. Total study duration is up to 186 days (~6 months) including an up to 18 day Screening period. Participants will be evaluated for safety, tolerability and efficacy bi-weekly during the first 4 weeks of treatment, and thereafter every 4 weeks for the duration of the study. Pharmacokinetics (PK) of Arikayce™ in blood, sputum and 24-hour urine will be determined in a subgroup of study participants who consent to PK evaluation.

At the completion of the TR02-108 protocol, participants who have consented and meet study safety criteria may enroll in the long-term, open-label, multi-cycle extension study of 590 mg of Arikayce™ (under a separate protocol TR02-110). Arikace™, Arikayce™, Liposomal Amikacin for Inhalation (LAI), and Amikacin Liposome Inhalation Suspension (ALIS) may be used interchangeably throughout this study and other studies evaluating amikacin liposome inhalation suspension.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent or assent
* Confirmed diagnosis of CF
* History of chronic infection with Pseudomonas aeruginosa
* Sputum culture positive for Pseudomonas aeruginosa at Screening
* FEV1 ≥ 25% of predicted value at Screening

Key Exclusion Criteria:

* FEV1 <25% of predicted at Screening
* History of major complications of lung disease within 8 weeks prior to Screening
* Hemoptysis of ≥60 mL in a 24-hour period within 4 weeks prior to Screening
* History of positive culture for Burkholderia cepacia within 2 years prior to Screening
* History of pulmonary tuberculosis or non-tuberculous mycobacterial lung disease treated within 2 years prior to Screening or requiring treatment at the time of screening
* History of Allergic Broncho-Pulmonary Aspergillosis or any other condition requiring systemic steroids at a dose ≥ equivalent of 10 mg/day of prednisone within 3 months prior to Screening
* Presence of any clinically significant cardiac disease
* History of lung transplantation
* Daily, continuous oxygen supplementation or nighttime supplemental oxygen requirement of greater than 2 L/min
* Administration of any investigational products within 8 weeks prior to study Day 1
* Smoking tobacco or any substance within 6 months prior to screening or anticipated inability to refrain from smoking throughout the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2012-02-29 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Eagle, MD, Study Director — Insmed Incorporated
Locations (62):
- Vienna, Austria
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Bulgaria (4):
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
- Canada (3):
  - Hamilton, Ontario
  - Halifax
  - Vancouver
- Copenhagen, Denmark
- France (7):
  - Bron
  - Lille
  - Montpellier
  - Nancy
  - Paris
  - Pierre-Bénite
  - Rouen
- Germany (6):
  - Berlin
  - Essen
  - Hamburg
  - Hanover
  - Kiel
  - München
- Greece (2):
  - Athens
  - Marousi
- Hungary (3):
  - Budapest
  - Debrecen
  - Szeged
- Dublin, Ireland
- Italy (8):
  - Ancona
  - Brescia
  - Catania
  - Genova
  - Milan
  - Parma
  - Roma
  - Verona
- Utrecht, Netherlands
- Poland (7):
  - Gdansk
  - Lodz
  - Lublin
  - Poznan
  - Rabka-Zdrój
  - Rzeszów
  - Warsaw
- New Belgrade, Serbia
- Slovakia (3):
  - Banská Bystrica
  - Bratislava
  - Košice
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia
- Gothenburg, Sweden
- United Kingdom (7):
  - Birmingham
  - Glasgow
  - Leeds
  - Liverpool
  - London
  - Nottingham
  - Penarth

REFERENCES:
- [Derived] Bilton D, Pressler T, Fajac I, Clancy JP, Sands D, Minic P, Cipolli M, Galeva I, Sole A, Quittner AL, Liu K, McGinnis JP 2nd, Eagle G, Gupta R, Konstan MW; CLEAR-108 Study Group. Amikacin liposome inhalation suspension for chronic Pseudomonas aeruginosa infection in cystic fibrosis. J Cyst Fibros. 2020 Mar;19(2):284-291. doi: 10.1016/j.jcf.2019.08.001. Epub 2019 Aug 23. PMID 31451351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 302 participants were randomized. 8 were not treated.
Groups:
- Arikayce™: Arikayce™ is liposomal amikacin for inhalation
  Liposomal amikacin for inhalation (Arikayce™) using the PARI Investigational eFlow® Nebulizer: Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * Liposomal amikacin for inhalation will be administered for 3 cycles where each cycle consists of 28 days on-treatment followed by 28 days off-treatment.
- TOBI®: TOBI® is tobramycin inhalation solution
  Tobramycin inhalation solution using a PARI LC® Plus nebulizer: 300 mg tobramycin inhalation solution is administered twice a day using a PARI LC® Plus nebulizer.
  * Nebulization time is approximately 20 minutes for each administration.
  * Tobramycin inhalation solution will be administered for 3 cycles where each cycle consists of 28 days on-treatment followed by 28 days off-treatment
Period: Overall Study
Arm/Group | Arikayce™ | TOBI®
Started (Number of participants treated) | 148 | 146
Completed | 134 | 140
Not Completed | 14 | 6
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — similar reason to those listed above | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arikayce™ | TOBI® | Total
Number analyzed (Participants) | 148 | 146 | 294
Age, Customized [Count of Participants; unit: Participants] — Population: Modified intent-to-treat (mITT; received at least 1 dose of study drug)
  Participants
    Age: 6-12 years | 27 | 26 | 53
    Age: >12-18 years | 34 | 33 | 67
    Age: >18 years | 87 | 87 | 174
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Modified intent-to-treat (mITT; received at least 1 dose of study drug)
  Participants
    Female | 69 | 70 | 139
    Male | 79 | 76 | 155
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — In TOBI arm , one patient was not recorded for ethnicity. Population: Modified intent-to-treat (mITT; received at least 1 dose of study drug)
  Participants
    Ethnicity: number analyzed (Participants) | 148 | 145 | 293
    Ethnicity: Caucasian | 139 | 141 | 280
    Ethnicity: Hispanic | 5 | 3 | 8
    Ethnicity: African | 1 | 0 | 1
    Ethnicity: Other | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Function Test: Forced Expiratory Volume in 1 Second (FEV1)
Description: Relative Change (%) from baseline to end of study (Day 168) in FEV1 (1 second)
Time Frame: Baseline to168 days
Population: The PP is the primary analysis population for the primary efficacy analysis
Measure: Mean (Standard Deviation); unit: Percent (%) change
Arm/Group | Arikayce™ | TOBI®
Number analyzed (Participants) | 129 | 137
Percent (%) change | 0.47 (13.930) | 1.67 (16.050)

2. Secondary Outcome: Pumonary Function Test: Forced Expiratory Volume in 1 Second (FEV1)
Description: Relative changes (%) from baseline to Study Days 14, 28, 57, 84, 113, 140, 168 in FEV1
Time Frame: Baseline, Day 14, Day 28, Day 57, Day 84, Day 113, Day 140 and Day 168.
Population: Modified intent-to-treat (mITT; received at least 1 dose of study drug)
Measure: Mean (Standard Deviation); unit: percentage (%) change
Arm/Group | Arikayce™ | TOBI®
Number analyzed (Participants) | 148 | 146
percentage (%) change
  Day 14: number analyzed (Participants) | 142 | 131
  Day 14 | 2.59 (13.332) | 6.64 (15.669)
  Day 28: number analyzed (Participants) | 114 | 114
  Day 28 | 0.79 (14.745) | 3.32 (14.715)
  Day 57: number analyzed (Participants) | 132 | 131
  Day 57 | -3.49 (12.319) | 0.70 (14.510)
  Day 84: number analyzed (Participants) | 110 | 104
  Day 84 | 0.44 (14.350) | 3.59 (14.642)
  Day 113: number analyzed (Participants) | 127 | 132
  Day 113 | -0.90 (12.028) | 0.42 (14.434)
  Day 140: number analyzed (Participants) | 103 | 105
  Day 140 | 0.43 (15.299) | 1.37 (16.563)
  Day 168: number analyzed (Participants) | 133 | 137
  Day 168 | -0.12 (14.326) | 1.58 (15.970)

3. Secondary Outcome: Number of Participants Experiencing a Pulmonary Exacerbation
Description: Number of participants experiencing a pulmonary exacerbation measured by number with event and number censored
Time Frame: 168 days
Population: Modified intent-to-treat (mITT; received at least 1 dose of study drug)
Measure: Number; unit: participants
Arm/Group | Arikayce™ | TOBI®
Number analyzed (Participants) | 148 | 146
participants
  Number with Event | 73 | 63
  Number Censored | 75 | 83
Statistical Analysis 1: Comparison: Arikayce™ vs TOBI®; Stratified Cox proportional hazards model; Test type: Superiority; p = 0.0286, Regression, Cox; Cox Proportional Hazard = 1.51, 95% CI 2-sided [1.07 to 2.13]

4. Secondary Outcome: Number of Participants to First Antipseudomonal Antibiotic Treatment for Pulmonary Exacerbation
Description: Number of participants to first antipseudomonal antibiotic treatment for pulmonary exacerbation measured by number with event and number censored
Time Frame: 168 days
Population: Modified intent-to-treat (mITT; received at least 1 dose of study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | Arikayce™ | TOBI®
Number analyzed (Participants) | 148 | 146
Participants
  Number with Event | 55 | 48
  Number Censored | 93 | 98
Statistical Analysis 1: Comparison: Arikayce™ vs TOBI®; Test type: Superiority; p = 0.6031, Regression, Cox; Cox Proportional Hazard = 1.12, 95% CI 2-sided [0.76 to 1.66]

5. Secondary Outcome: Number of Participants to First All Cause Hospitalization
Description: Number of participants to first all cause hospitalization measured by number with event and number censored
Time Frame: 168 days
Population: Modified intent-to-treat (mITT; received at least 1 dose of study drug)
Measure: Number; unit: participants
Arm/Group | Arikayce™ | TOBI®
Number analyzed (Participants) | 148 | 146
participants
  Number with Event | 24 | 29
  Number Censored | 124 | 117
Statistical Analysis 1: Comparison: Arikayce™ vs TOBI®; Test type: Superiority; p = 0.4861, Regression, Cox; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.49 to 1.44]

6. Secondary Outcome: Change in Density (Log CFU) in Pseudomonas Aeruginosa in Sputum
Description: Change in density (Log CFU) from baseline in Pseudomonas aeruginosa in sputum
Time Frame: Baseline, Day 14, Day 28, Day 57, Day 84, Day 113, Day 140 and Day 168
Population: Modified intent-to-treat (mITT; received at least 1 dose of study drug)
Measure: Mean (Standard Deviation); unit: Log 10 CFU
Arm/Group | Arikayce™ | TOBI®
Number analyzed (Participants) | 148 | 146
Log 10 CFU
  Baseline: number analyzed (Participants) | 134 | 131
  Baseline | 6.872 (1.8806) | 6.510 (2.3202)
  14 days: number analyzed (Participants) | 131 | 120
  14 days | -1.124 (2.0542) | -1.663 (2.4017)
  28 days: number analyzed (Participants) | 129 | 120
  28 days | -1.208 (2.1594) | -1.453 (2.4440)
  57 days: number analyzed (Participants) | 122 | 120
  57 days | -0.210 (1.9874) | -0.098 (1.7446)
  84 days: number analyzed (Participants) | 120 | 119
  84 days | -0.945 (2.2223) | -1.182 (2.6914)
  113 days: number analyzed (Participants) | 114 | 118
  113 days | -0.613 (2.1928) | -0.135 (2.3461)
  140 days: number analyzed (Participants) | 117 | 116
  140 days | -1.440 (2.4357) | -1.315 (2.2300)
  168 days: number analyzed (Participants) | 117 | 118
  168 days | -0.725 (2.0073) | -0.136 (2.1750)

7. Secondary Outcome: Relative Percent (%) Change in Respiratory Symptoms as Measured by the CFQ-R
Description: Quality of Life was measured by the absolute change from baseline in the Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory scale. Disease specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms in patients with a diagnosis of cystic fibrosis. Scores range from 0 to 100, with higher scores indicating better health. Scores for each Health Related Quality of Life (HRQoL) domain; after recoding, each item is summed to generate a domain score and standardized.
Time Frame: Day 14, Day 28, Day 57, Day 84, Day 113, Day 140 and Day 168
Population: Modified intent-to-treat (mITT; received at least 1 dose of study drug)
Measure: Least Squares Mean (Standard Error); unit: Percent (%) change
Arm/Group | Arikayce™ | TOBI®
Number analyzed (Participants) | 148 | 146
Percent (%) change
  Day 14: number analyzed (Participants) | 141 | 136
  Day 14 | 13.65 (2.995) | 8.81 (3.019)
  Day 28: number analyzed (Participants) | 143 | 138
  Day 28 | 15.54 (3.363) | 11.03 (3.419)
  Day 57: number analyzed (Participants) | 137 | 134
  Day 57 | 8.00 (3.120) | 7.97 (3.146)
  Day 84: number analyzed (Participants) | 136 | 135
  Day 84 | 13.20 (3.079) | 8.55 (3.111)
  Day 113: number analyzed (Participants) | 131 | 135
  Day 113 | 3.58 (3.323) | 5.03 (3.290)
  Day 140: number analyzed (Participants) | 130 | 135
  Day 140 | 13.84 (3.060) | 6.10 (3.079)
  Day 168: number analyzed (Participants) | 128 | 131
  Day 168 | 12.06 (3.784) | 8.07 (3.790)

ADVERSE EVENTS:
Arm/Group | Arikayce™ | TOBI®
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/146
Serious Adverse Events (participants affected / at risk) | 26/148 | 29/146
Other Adverse Events (participants affected / at risk) | 114/148 | 91/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arikayce™ (N=148) | TOBI® (N=146)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 24 (28) | 23 (28)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0)
Pulmonary function test decreased (Investigations) | 0 (0) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arikayce™ (N=148) | TOBI® (N=146)
diarrhoea (Gastrointestinal disorders) | 10 (12) | 5 (5)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 82 (138) | 72 (117)
Nasopharyngitis (Infections and infestations) | 24 (29) | 33 (43)
Upper respiratory tract infection (Infections and infestations) | 15 (21) | 9 (14)
Rhinitis (Infections and infestations) | 9 (10) | 9 (9)
Headache (Nervous system disorders) | 12 (22) | 5 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 24 (53) | 10 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 11 (24)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 (28) | 8 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 6 (7)
General disorders (General disorders) | 20 (23) | 10 (13)
Investigations (Investigations) | 12 (15) | 10 (11)
Musculoskeletal and connective (Musculoskeletal and connective tissue disorders) | 12 (14) | 10 (12)
Skin and subcutaneous (Skin and subcutaneous tissue disorders) | 8 (10) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the signed Investigator Agreement in the study protocol and protocol amendments, the PI agreed "not to originate or use the name of Insmed Incorporated, or study drug code in any publicity, news release, or other public announcement, written or oral, whether to the public, press, or otherwise, relating to this protocol, to any amendment to the protocol, or to the performance of this protocol, without the prior written consent of Insmed Incorporated."